CLINICAL TRIAL: NCT02719678
Title: Epidemiological Studies of Health Effects of General Examinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Allan Linneberg, Professor, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Monica Intervention
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Invitation to up to three general health checks over a 10-year period
  Interventions: Other: General health checks
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: General health checks — The intervention group is invited to up to three general health checks over a 10-year period
  Arms: Intervention group

SUMMARY:
The effect of systematic health examinations and screening of the general population is under debate. Recently, a large Danish randomized study found that systematic screening of risk factors and lifestyle advice in the general population did not have a preventive effect on coronary heart disease, stroke or all-cause mortality. However, there are still very few completed randomized studies, and the effect on other diseases remains unclear. The purpose is to investigate whether repeated health examinations with screening of various risk factors in an unselected population prevent long-term incidence of ischemic heart disease, stroke, total and cause-specific mortality, diabetes, dementia, chronic obstructive pulmonary disease and various forms of cancer. A preliminary protocol was submitted and approved by the Danish Data Protection Agency before the registry-based data on primary and secondary outcomes were received by the investigator.

DETAILED DESCRIPTION:
Introduction The effect of systematic health examinations and screening of the general population is under debate. Recently, a large Danish randomized study found that systematic screening of risk factors and lifestyle advice in the general population did not have a preventive effect on coronary heart disease, stroke or all-cause mortality. However, there are still very few completed randomized studies, and the effect on other diseases remains unclear.

Purpose The purpose is to investigate whether repeated health examinations with screening of various risk factors in an unselected population prevent long-term incidence of ischemic heart disease, stroke, total and cause-specific mortality, diabetes, dementia, chronic obstructive pulmonary disease and various forms of cancer.

Research question Can health examinations with screening of various risk factors prevent the long-term incidence of ischemic heart disease, stroke, total and cause-specific mortality, diabetes, dementia, chronic obstructive pulmonary disease and various forms of cancer?

Data and method For the Danish Monica1 study, a random sample of the general population (adults) in Copenhagen County in 1982 and 1983 was extracted, consisting of a total of 17,845 people. These individuals were randomly divided into two groups, one group was offered a general medical examination while participating in the study, while the control group was not invited and remained unaware of the intervention. The intervention was thus an examination with measuring of e.g., blood pressure, cholesterol level and body mass index as well as subsequent conversation with a nurse. Participants were invited 3 times at 5-year intervals. Data from the intervention group (4,807 people) and the control group (13,038 persons) will be linked to register data from the Danish Civil Registration Register, the Cause of Death Register, the National Patient Register, the Diabetes Register and the Cancer Register. The effect of the intervention will be examined using Cox regression with intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* age 30, 40, 50 or 60 years
* living in one of the pre-specified municipalities of Copenhagen

Exclusion Criteria:

* none

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17845 (Actual)
Dates: Start 1982-01; Primary Completion 1984-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
cardiovascular disease | 30 years of follow-up
all-cause mortality | 30 years of follow-up

SECONDARY OUTCOMES:
cancer | 30 years of follow-up
Diabetes | 30 years of follow-up
COPD | 30 years of follow-up
Tobacco-related diseases | 30 years of follow-up
Dementia | 30 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Allan Linneberg, Principal Investigator — Research Centre for Prevention and Health
Locations (1):
- Research Centre for Prevention and Health, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon request and approval from the Ethics Committee.